CLINICAL TRIAL: NCT00366132
Title: DermaGold Indicated for Use of Shockwave Treat of Diabetic Foot Ulcers in Patients With Diabetes Mellitus
Brief Title: Safety & Efficacy Study for the Use of Extracorporeal Shockwaves in the Treatment of Diabetic Foot Ulcers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tissue Regeneration Technologies (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G050198
Record Dates: First submitted 2006-08-17; First posted 2006-08-18 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Chronic Diabetic Foot Ulcers
Keywords: Diabetic; Foot Ulcers; TRT; DermaGold; Shockwave; ESWT; Diabetes Mellitus
MeSH Terms: conditions — Foot Ulcer; Diabetes Mellitus

INTERVENTIONS:
Device: Extracorporeal Shockwaves

SUMMARY:
The purpose of this clinical study is to compare the safety and effectiveness of shockwave treatment combined with standard-of-care treatment, to standard-of-care treatment alone to induce healing of a chronic plantar foot ulcer in subjects with diabetes mellitus. For the purpose of this study, the definition of plantar foot ulcer is a wound or open sore that involves the plantar(bottom) aspect of the foot, and the definition of chronic is a duration of 6 weeks or greater with a lack of response to treatment.

DETAILED DESCRIPTION:
Diabetic foot complications are the most common cause of nontraumatic lower extremity amputations in the industrialized world. The risk of lower extremity amputation ranges from 15 to 46 times higher in diabetics than in persons who do not have diabetes mellitus. Furthermore, foot complications are the most frequent reason for hospitalization in patients with diabetes, accounting for up to 25 percent of all diabetic admissions in the United States and Great Britain. The vast majority of diabetic foot complications resulting in amputation begin with the formation of skin ulcers. Early detection and appropriate treatment of these ulcers may prevent up to 85 percent of amputations. (Armstrong)

The primary goal in the treatment of diabetic foot ulcers is to obtain wound closure. Rest, elevation of the affected foot, and relief of pressure are basic treatments that are usually initiated when the patient first presents with a foot ulcer. A postoperative shoe or another type of pressure-relieving footwear is also often prescribed. Crutches or a wheelchair might also be recommended to totally off-load pressure from the foot. Necrotic tissue is debrided to allow full visualization of the extent of the ulcer, to allow detect underlying abscesses or sinuses, and to support healing. Wet-to-wet dressings are used to provide a warm, moist environment that is protected from external contamination is most conducive to wound healing. Additional options include numerous topical medications and gels, and special dressings, including semipermeable films, foams, hydrocolloids, and calcium alginate swabs.

When these more conservative treatments fail, another recently developed nonoperative option is available. The genetically engineered platelet-derived growth factor becaplermin (Regranex Gel, OMJ Pharmaceuticals, Inc.) is approved for use on neuropathic diabetic foot ulcers and can expedite healing. Growth factors stimulate chemotaxis and mitogenesis of neutrophils, fibroblasts, and monocytes, as well as other components that form the cellular basis of wound healing.

When nonoperative treatments fail, skin grafting is often required to achieve wound closure. In addition to autologous donor tissue for the graft procedure, bioengineered skin (Apligraf, Organogenesis, P950032/S016) and human dermis (Dermagraft, Smith & Nephew, P000036) are new types of biologically active implants approved for diabetic foot ulcers that are derived from fibroblasts of neonatal foreskins. These bioengineered products enhance healing by acting as delivery systems for growth factors and extracellular matrix components through the activity of live human fibroblasts contained in their dermal elements. (Frykberg)

Despite the variety of modalities available to treat diabetic foot ulcers, the US Center for Disease Control reports that the age-adjusted lower extremity amputation rate for persons with diabetes is 5.5 per 1,000 persons with diabetes, which is was 28 times that of persons without diabetes.

ESWT for Soft Tissue Indications

The use of extracorporeal shock waves for clinical applications was introduced in the United States more than 20 years ago; the first indication for use approved by FDA was for treatment of renal calculi (kideny stones). Since that time, the clinical applications of extracorporeal shock wave therapy (ESWT) have been expanded to include treatment of chronic proximal plantar fasciitis (P990086, HealthTronics OssaTron; P000048, Dornier EPOS Ultra; P040026, Orthospec Extracorporeal Shock Wave Device; P040039, Orthometrix Orbasone Pain Relief System) and chronic lateral epicondylitis (P990086/S003, HealthTronics OssaTron; P010039, Siemens Sonocur Basic). In addition, there are numerous reports in the clinical and pre-clinical literature of shockwave therapy used to treat orthopedic conditions such as fracture non-unions, femoral head necrosis, and non-orthopedic conditions related to tissue healing.

Treatment with extracorporeal shock waves has been shown to be associated with neovascularization in an animal model. Further, since several shockwave systems have been approved through the PMA process for treatment of chronic proximal plantar fasciitis and chronic lateral epicondylitis, there is a large amount of data regarding the safety of these devices in treating soft tissue. The research done by Meirer et al. (2005) and by Nishida et al. (2004) suggests that local delivery of shockwave therapy results in increased release of growth factors and improved circulation in the wound.

Because of the promising association between ESWT and tissue healing, the favorable risk / benefit profile of the devices approved for treatment of soft tissue indications, and the European clinical experience with ESWT for wound healing, it is hypothesized that extracorporeal shock wave treatment (ESWT) could be beneficial in treating diabetic foot ulcers. Therefore, this IDE describes a clinical study designed to determine the safety and effectiveness of the DermaGold® ESW System when used to induce healing of chronic plantar foot ulcers in patients with diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a single chronic plantar foot ulcer that has persisted for a minimum of 6 weeks duration
* History of Type 2 diabetes mellitus; (track/ask if insulin dependent)
* Capable of wound care at home;
* The ulcer measures > 1 cm and <4 cm at any dimension
* The ulcer is Stage 1 or 2A according to the classification system described by Lavery et al.
* Stage 1 - superficial wounds through the epidemis or epidermis and dermis that did not penetrate to tendon, capsule or bone.
* Stage 2A - Clean wounds that penetrated to tendon or capsule.
* Palpable pedal pulse in the affected leg OR peripheral vascular disease evaluation demonstrating acceptable blood supply to affected foot;
* Subjects age > 18 years;
* The Investigator has completed a medical history and a physical examination to assure that the subject meets all study enrollment criteria;
* The subject is willing and able to read, understand and sign the study specific informed consent form; and
* The subject agrees to comply with study protocol requirements, including the shockwave procedure, self-care of the wound (e.g., wet to wet dressings, orthotics) and all follow up visit requirements.

Exclusion Criteria:

* Pregnancy
* Type I diabetes
* Plantar foot ulcer extends to and /or involves the bone or joint;
* Ulcers are present on both feet
* Multiple ulcers on the foot
* Clinical evidence of cellulitis at the ulcer site or surrounding area;
* Ulcers that have purulent exudates or malodorous exudates on visual examination
* Diagnosis of a chronic plantar foot ulcer that has persisted for >1 year.
* Peripheral vascular disease per the study enrollment work-up requiring vascular surgery intervention.
* ABI (Ankle Brachial Index) < 0.6 Ulcer debridement under anesthesia in OR required within the 2 week observation phase,
* Lower extremity revascularization procedure (e.g. PTA, graft, etc.) within eight (8) weeks of the study screening visit.
* Uncorrected biomechanical abnormalities that cause or contribute to the affected lower extremity ulcer; (e.g. tight Achilles tendon, hammer toe, Charcot foot etc.)
* Surgical procedure to correct biomechanical abnormities (e.g., lengthening of the Achilles tendon. correction of hammer toe, Charcot foot correction) within eight (8) weeks of the study screening visit;
* Deep vein thrombosis within 6 months of study screening visit;
* Clinical evidence of lymphadema;
* Active or previous (within 60 days prior to the study screening visit) chemotherapy;
* Treatment of the plantar foot ulcer with growth factors, prostaglandin therapy or vasodilator therapy during the 2 week observation phase.
* Subject on steroid therapy
* Sickle cell anemia
* Infection with Human Immunodeficiency Virus
* Immunodeficiency disorders
* Severe protein malnutrition - serum albumin < 2.0g/dl
* Severe anemia - Hgb < 7 g/dl (males) or < 6.5 (females)
* Recent treatment (within 60 days prior to the study screening visit) with immunosuppresants, radiation, or biologically active cellular / acellular products;
* Current history of substance abuse.
* Physical or mental disability or geographical concerns (residence not within reasonable travel distance) that would hamper compliance with required study visits;
* Current participation in another clinical investigation of a medical device or a drug, or recent participation in such a study within 30 days prior to study enrollment; or
* The Investigator believes that the subject will be unwilling or unable to comply with study protocol requirements, including the shock wave treatment procedure, standard-of-care self-care requirements, and all study-related follow up visit requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2006-03

PRIMARY OUTCOMES:
Time to Complete Wound Healing

SECONDARY OUTCOMES:
o A comparison of the total number of subjects with a final status of "Healed" in the active versus control group
o Partial healing at 12 weeks post treatment ((size of wound compared to baseline));
o Results of quantitative wound cultures (Ulcers with a quantitative wound culture with a bacterial count greater than 105 per gram of tissue will be defined as an infected ulcer);
o The percentage of the wound that has healed
o The number of shock wave treatments performed
o Durability of wound closure (i.e., status of wound at one week following determination of "healed")

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Calvary Hospital, The Bronx, New York
  - Akron General, Akron, Ohio
  - University of Texas Medical Branch, Galveston, Texas
  - Podiatry Group of South Texas, San Antonio, Texas